CLINICAL TRIAL: NCT06247306
Title: Probing the Influence of Neural Stress Responses on Problematic Alcohol Use With Real-time fMRI Neurofeedback (C04)
Brief Title: Using Neurofeedback to Understand the Relationship Between Stress and Alcohol Consumption
Acronym: NeuStress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: U1111-1302-2402; TRR265-C04 (Other: Deutsche Forschungsgemeinschaft)
Record Dates: First submitted 2024-01-13; First posted 2024-02-07 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Alcohol Abuse; Craving; Psychosocial Stressor; Neural Stress Response
Keywords: functional Magnetic Resonance Imaging (fMRI); psychosocial stress; real-time fMRI neurofeedback (rtfMRI neurofeedback); problematic alcohol use; cortisol; Ecological momentary assessment (EMA)
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Firstly,.all participants are assigned to either the experimental or the sham-control (Yoke-control) group through a fully automated, double-blind procedure. All participants undergo one neurofeedback (NFB) session with two runs à 9:30 mins. The NFB runs have a block structure with alternating periods/ blocks of self-regulation and rest. Participants of both groups receive the instruction to decrease their stress-response (thus, upregulating their ACC activity), through whichever strategy helps them to achieve this goal. The experimental group receives real-time fMRI feedback of their respective ACC activity. The sham-control group or Yoke-control group receives a previously acquired recording of the neurofeedback signal from a different participant instead of their own real-time ACC activity.
Who Masked: Participant, Investigator
Masking Description: Next to the investigator and participants, research assistants as well as medical technical radiology assistants (MTRAs) will be blinded to the conditions. Only after the 6-week long ecological momentary assessment is completed are participants as well as investigators, MTRAs and research assistants debriefed concerning the participants group assignment (experimental or Yoke-control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real-time fMRI neurofeedback (of the ACC) (Experimental): Participants are instructed to reduce their stress-response by attempts to upregulate the ACC activity contigent on real-time feedback.
  Interventions: Behavioral: ScanSTRESS fMRI-paradigm (Streit et al., 2014); Behavioral: real-time fMRI neurofeedback
- Yoke-control group (Sham Comparator): Participants receive previously recorded feedback signal from other participants' ACC activity instead of their own live ACC activity.
  Interventions: Behavioral: ScanSTRESS fMRI-paradigm (Streit et al., 2014); Behavioral: real-time fMRI neurofeedback

INTERVENTIONS:
Behavioral: ScanSTRESS fMRI-paradigm (Streit et al., 2014) — The task is conducted within the MRI scanner and consists of two runs each lasting 11:20 mins., employs a block design and has two different conditions (performance, relaxation), as well as two different task within each condition. Participants undergo the following 2 tasks during the performance condition under time pressure: 1) serial subtraction, 2) a figure matching task. During the performance condition, all participants receive feedback (work faster, mistake, too slow) and are reprimanded concerning their performance. Two investigators in white coats observe the participants with critical facial expression, which is projected to participants through live-video feed during the tasks. The relaxation condition includes easy versions of arithmetic and figure matching task without time constrains or any type feedback on their performance. Performance and relaxation phases are appear in alternating order.
Behavioral: real-time fMRI neurofeedback — Two real-time fMRI neurofeedback sessions of 9:30 minutes each are conducted. During these sessions, the participants are instructed to regulate a feedback signal from the ACC. Participants are assigned to either the experimental or Yoke-control group through an automated double-blind procedure. In the neurofeedback sessions, participants in the experimental group receive a feedback signal indicating their current ACC activation. Participants in the control group receive the recorded feedback signal from another participant. The neurofeedback sessions follow a block structure with alternating feedback and rest periods.
  Before, between, and after the two sections of the fMRI examination, subjective stress levels and alcohol craving are assessed, and saliva samples are collected for cortisol level determination.

SUMMARY:
In this research project, the aim is to discover the role specific brain networks play in the relationship between stress reactions and the desire for alcohol and alcohol consumption. To investigate this question, various brain imaging methods as well as cognitive tasks are combined. Various questionnaires are sampled and brain scans are conducted.

Individuals interested in participating in the study have to fulfill certain criteria...

* no serious medical or mental health diagnosis
* problematic alcohol drinking habits
* interested in improving drinking habits

  ...and undergo various non-invasive procedures
* filling out several questionnaires concerning personality and habits
* undergoing a mental performance task while being in a brain scanner (MRI)
* attempting to regulate their own brain activity while lying in the MRI scanner
* filling out an electronic diary for 6 weeks - concerning daily mood, stress, and alcohol habits

Participants will be randomly allocated to either one of 2 experimental groups. Both groups undergo the same tasks, receive the same instructions and only differ regarding some aspects of the brain self-regulation task .

DETAILED DESCRIPTION:
While it is well known and long acknowledged in scientific research that stress and alcohol consumption are closely linked, the actual relationship is complex, and the underlying mechanisms are only partially understood. To investigate the effects of acute stress under controlled conditions, experimental procedures, stress tests, and related paradigms are often employed. Studies on alcohol addiction generally indicate an increase in acute cravings following the experimental induction of stress. Neurologically, acute stress induction is associated with activation changes in widespread networks. In particular, research employing stress tests found increased activations in striatum, thalamus and limbic areas and deactivations in anterior cingulate cortex (ACC) as well as ventromedial prefrontal cortex (vmPFC), areas often associated with emotion regulation during stress induction. Given their role in emotion regulation, deactivations in these areas could reflect a reduction in emotional control during acute stress. Deactivation of these areas during experimentally induced stress has also been linked to problematic alcohol consumption and increased alcohol cravings.

This study aims to elucidate how neurocognitive processes during stress influence alcohol cravings and consumption. To this end, participants with problematic alcohol consumption will be recruited. After having filled out various questionnaires pertaining to their biographical data, alcohol consumption and personality traits, participants will be experimentally stressed during a brain scan using functional Magnetic Resonance Imaging (fMRI). To reliably induce psychosocial stress, the ScanSTRESS test, a paradigm explicitly conceptualized for usage during MRI scanning, will be employed. Once the stress test is completed, participants will attempt to regulate their own neurological stress response through upregulation of the ACC using information about their current stress-induced brain activity (neurofeedback). Additionally, saliva samples will be regularly taken during the experiment to biologically observe the stress response through cortisol measurements. This will be followed by a 6-week follow-up phase, during which participants will be specifically asked about their alcohol cravings, alcohol consumption, and daily stress experiences.

By employing real-time fMRI neurofeedback, this study creates experimental conditions in which participants can self-regulate the neural stress response of the targeted brain network. Nonspecific effects of the neurofeedback paradigm are controlled using a sham condition (Yoke-control group). Participants are randomly assigned to either the control group or the real neurofeedback group (experimental group). This approach allows for the investigation of the neural self-regulation abilities of emotional control networks and their role in the connection between stress, alcohol cravings, and drinking behavior in real life.

In summary, this study aims to examine the relationship between the self-regulation abilities of neural stress responses and real-life drinking behavior.

Investigators hypothesize that 1) the stress experiment significantly increases acute self-reported stress in participants, 2) specifically stress-induced patterns of neural activity, namely increased striatal and thalamic activity as well as decreased ACC activity, predict alcohol cravings and consumption, 3) the experimental neurofeedback group exhibits higher ACC activity during brain self-regulation than the control group, 4) the experimental group shows lower alcohol craving/consumption during the follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Presence of 2 to a maximum of 5 criteria for alcohol use disorder according to DSM-5
* no clinical necessity for detoxification treatment
* participants may have a moderate cannabis use disorder and tobacco use disorder
* Capacity for consent and ability to use self-assessment scales
* Sufficient knowledge of German
* Willingness to use a mobile phone with Android operating system

Exclusion Criteria:

* Lifetime diagnosis of bipolar or psychotic disorder or a substance use disorder according to Diagnostical and Statistical Manual of Mental Disorders - 5 (DSM-5) that is not alcohol, cannabis, or tobacco use disorder
* Current substance use other than cannabis and tobacco
* Current diagnosis of one of the following conditions according to DSM-5: (hypo)manic episode, major depression, generalized anxiety disorder, post-traumatic stress disorder, borderline personality disorder, or obsessive-compulsive disorder
* History of severe head trauma or other severe central neurological disorders (dementia, Parkinson&#39;s disease, multiple sclerosis)
* Pregnancy or lactation
* Use of medications known to interact with the central nervous system within the last 10 days; testing at least four half-lives after the last dose
* Exercising the prerogative of the &#34;Right not to know&#34; in the context of incidental findings during an examination or investigation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Neurofeedback/Stress-Regulation Parameters | Assessed during each of the two neurofeedback runs, 9:30 minutes respectively
  During neurofeedback runs, participants' activation changes in the region of interest (ROI) is sampled and compared to a previously determined baseline activation (localizer task). The ROI participants are tasked to regulate is the ACC. Successful regulation is characterized as significant increase (upregulation) of the ACC as compared to baseline activation.
Stress-induced neural activation | 23 minutes - 2 runs lasting 11:20 minutes each
  Regional activation and network activation characterized during ScanSTRESS paradigm through means of contrast testing ("performance" condition vs "rest" condition)
Cortisol | Three measurement time points: 1. T0: 10 minutes before the ScanStress Test 2. T1: 33 minutes after T0 (after the ScanStress Test) 3. T2: 52 minutes after T0 (after both fMRI paradigms -ScanStress & Neurofeedback)
  Cortisol will be assessed through saliva samples
Craving | Three measurement time points: 1. T0: 10 minutes before the ScanStress Test 2. T1: 33 minutes after T0 (after the ScanStress Test) 3. T2: 52 minutes after T0 (after both fMRI paradigms -ScanStress & Neurofeedback)
  Self-report assessment questionnaire, Craving Automated Scale for Alcohol (CAS-A, Vollstädt-Klein et. al., 2015),
Ecological/electronic Momentary Assessment (movisensXS) | 6 weeks starting from the conclusion of the neurofeedback intervention
  Participants install the study app (movisensXS) on their mobile phones. During the six-week follow-up phase, data on daily stress experiences and alcohol consumption are collected through the study app. The study app assesses stress experiences, alcohol cravings, alcohol consumption, social interactions, health behavior, and coping with stress situations through short queries. The queries occur once daily at a random time between 10am and 8pm and last approximately 60 seconds. Participants can postpone the queries by up to 15 minutes or decline them altogether. Additionally, three extra queries regarding alcohol consumption are conducted once a week. During these queries, participants are asked to report their stress experiences, alcohol consumption, alcohol cravings, alcohol-related triggers, social interactions, coping with stress situations, health behavior (e.g., sleep duration), and goals related to alcohol consumption (duration of individual queries approx. 120 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Martin F Gerchen, PhD, Principal Investigator — Central Institute of Mental Health; Peter Kirsch, Prof., PhD, Principal Investigator — Central Institute of Mental Health; Falk Kiefer, MD, PhD, Principal Investigator — Central Institute of Mental Health
Locations (1):
- Central Institute of Mental Health - Department of Clinical Psychology, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
There will be collaborative data processing, sharing of data and storage of data at different locations as specified below.
  Research data will be stored on secure servers of the Center for Information Services and High-Performance Computing at the Dresden University of Technology (ZIH; Zellescher Weg 12, 01069 Dresden) and the ZI Mannheim. The data will be retained for 10 years after the completion or termination of the research project. Participants' data will be protected against unauthorized access, and anonymization will occur once the research purpose allows it. Data will be deleted at the latest after 10 years.
  Coding method: Double coding, access by project staff, emergency decoding possible during the project duration (MRT scans).
  Transfer of pseudonymized biomaterials/data to third parties: Name: Dresden University of Technology Address: Zellescher Weg 19, 01069 Dresden. There will be a transfer of pseudonymized saliva samples for cortisol level determination.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The biomaterials will be destroyed immediately after the completion of the work. All other data will become available at the start of the study and will be deleted 10 years after the completion of the study. Data sharing will not be possible 10 years after completion of the study.

REFERENCES:
- [Background] Wolkowicz NR, Peltier MR, Wemm S, MacLean RR. Subjective stress and alcohol use among young adult and adult drinkers: Systematic review of studies using Intensive Longitudinal Designs. Drug Alcohol Depend Rep. 2022 Mar 11;3:100039. doi: 10.1016/j.dadr.2022.100039. eCollection 2022 Jun. PMID 36845979
- [Background] Vollstadt-Klein S, Hermann D, Rabinstein J, Wichert S, Klein O, Ende G, Mann K. Increased activation of the ACC during a spatial working memory task in alcohol-dependence versus heavy social drinking. Alcohol Clin Exp Res. 2010 May;34(5):771-6. doi: 10.1111/j.1530-0277.2010.01149.x. Epub 2010 Mar 1. PMID 20201927
- [Background] Vollstadt-Klein S, Lemenager T, Jorde A, Kiefer F, Nakovics H. Development and validation of the craving automated scale for alcohol. Alcohol Clin Exp Res. 2015 Feb;39(2):333-42. doi: 10.1111/acer.12636. PMID 25684052
- [Background] Streit F, Haddad L, Paul T, Frank J, Schafer A, Nikitopoulos J, Akdeniz C, Lederbogen F, Treutlein J, Witt S, Meyer-Lindenberg A, Rietschel M, Kirsch P, Wust S. A functional variant in the neuropeptide S receptor 1 gene moderates the influence of urban upbringing on stress processing in the amygdala. Stress. 2014 Jul;17(4):352-61. doi: 10.3109/10253890.2014.921903. Epub 2014 Jun 16. PMID 24800784
- [Background] Sinha R, Li CS. Imaging stress- and cue-induced drug and alcohol craving: association with relapse and clinical implications. Drug Alcohol Rev. 2007 Jan;26(1):25-31. doi: 10.1080/09595230601036960. PMID 17364833
- [Background] Sinha R, Fox HC, Hong KA, Bergquist K, Bhagwagar Z, Siedlarz KM. Enhanced negative emotion and alcohol craving, and altered physiological responses following stress and cue exposure in alcohol dependent individuals. Neuropsychopharmacology. 2009 Apr;34(5):1198-208. doi: 10.1038/npp.2008.78. Epub 2008 Jun 18. PMID 18563062
- [Background] Seo D, Lacadie CM, Tuit K, Hong KI, Constable RT, Sinha R. Disrupted ventromedial prefrontal function, alcohol craving, and subsequent relapse risk. JAMA Psychiatry. 2013 Jul;70(7):727-39. doi: 10.1001/jamapsychiatry.2013.762. PMID 23636842
- [Background] Seo D, Lacadie CM, Sinha R. Neural Correlates and Connectivity Underlying Stress-Related Impulse Control Difficulties in Alcoholism. Alcohol Clin Exp Res. 2016 Sep;40(9):1884-94. doi: 10.1111/acer.13166. Epub 2016 Aug 8. PMID 27501356
- [Background] Koob GF, Le Moal M. Drug abuse: hedonic homeostatic dysregulation. Science. 1997 Oct 3;278(5335):52-8. doi: 10.1126/science.278.5335.52. PMID 9311926
- [Background] Kirschbaum C, Pirke KM, Hellhammer DH. The 'Trier Social Stress Test'--a tool for investigating psychobiological stress responses in a laboratory setting. Neuropsychobiology. 1993;28(1-2):76-81. doi: 10.1159/000119004. PMID 8255414
- [Background] Cox WM, Klinger E. A motivational model of alcohol use. J Abnorm Psychol. 1988 May;97(2):168-80. doi: 10.1037//0021-843x.97.2.168. No abstract available. PMID 3290306
- [Background] Clay JM, Parker MO. The role of stress-reactivity, stress-recovery and risky decision-making in psychosocial stress-induced alcohol consumption in social drinkers. Psychopharmacology (Berl). 2018 Nov;235(11):3243-3257. doi: 10.1007/s00213-018-5027-0. Epub 2018 Sep 12. PMID 30209533
- [Background] Clay JM, Adams C, Archer P, English M, Hyde A, Stafford LD, Parker MO. Psychosocial stress increases craving for alcohol in social drinkers: Effects of risk-taking. Drug Alcohol Depend. 2018 Apr 1;185:192-197. doi: 10.1016/j.drugalcdep.2017.12.021. Epub 2018 Feb 15. PMID 29462766
- [Background] Bush K, Kivlahan DR, McDonell MB, Fihn SD, Bradley KA. The AUDIT alcohol consumption questions (AUDIT-C): an effective brief screening test for problem drinking. Ambulatory Care Quality Improvement Project (ACQUIP). Alcohol Use Disorders Identification Test. Arch Intern Med. 1998 Sep 14;158(16):1789-95. doi: 10.1001/archinte.158.16.1789. PMID 9738608
- [Background] Blaine SK, Seo D, Sinha R. Peripheral and prefrontal stress system markers and risk of relapse in alcoholism. Addict Biol. 2017 Mar;22(2):468-478. doi: 10.1111/adb.12320. Epub 2015 Nov 5. PMID 26537217
- [Background] Amlung M, MacKillop J. Understanding the effects of stress and alcohol cues on motivation for alcohol via behavioral economics. Alcohol Clin Exp Res. 2014 Jun;38(6):1780-9. doi: 10.1111/acer.12423. Epub 2014 May 30. PMID 24890323